CLINICAL TRIAL: NCT00149331
Title: A Randomized Controlled Trial Comparing the Effects of Two Education Strategies About Insulin on Preferences and Perceptions About Insulin Therapy
Brief Title: The Effects of Two Education Strategies About Insulin on Patient Preferences and Perceptions About Insulin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 04-2429
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes, Insulin, Education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

INTERVENTIONS:
Behavioral: Structured education program

SUMMARY:
This study compared the impact of two educational strategies (an education program versus a pamphlet) on participants preferences for insulin and their perceptions about insulin and injections after attending an educational session with a diabetes educator about insulin.

Main research question: Among adults with type 2 diabetes who are potential candidates for insulin therapy, does an education strategy that involves a personal letter from the family physician, a presentation about insulin, and information about giving an injection, versus a pamphlet education strategy, effect: preference to accept insulin therapy; perceptions about insulin therapy; or perception about the injection?

DETAILED DESCRIPTION:
Many people with type 2 diabetes who need insulin therapy are often reluctant to start using insulin to manage their diabetes. This may be because they are worried about giving an injection and do not know enough about insulin to make an informed choice. This research is important because it will help researchers and health care providers better understand the feelings and educational support that patients need when they are thinking about starting insulin. This can help health care providers to better tailor the care they give to patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Have a diagnosis of type 2 diabetes mellitus in their medical chart
* Have suboptimal glycosylated hemoglobin (HgA1c > 7.5%) recorded in their chart as the most recent lab result
* Currently perform self-monitoring of blood glucose
* Able to understand written and spoken English

Exclusion Criteria:

* Are currently using, or have previously used insulin
* Have cognitive, visual, hearing or other medical impairment
* Have terminal malignancies or dementia
* Have psychiatric illness not controlled with medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86
Dates: Start 2005-07; Study Completion 2006-03

PRIMARY OUTCOMES:
Preference for Insulin therapy

SECONDARY OUTCOMES:
Perceptions about insulin therapy
Perceptions about injection
Satisfaction with the education session

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dolovich, PharmD MSc, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences - Henderson Site, Hamilton, Ontario, Canada